CLINICAL TRIAL: NCT06280599
Title: An Experimental Study of the Application of Transitional Care Model on Patients With Stroke
Brief Title: Transitional Care Model for Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Ita Daryanti Saragih, Principal Investigator, Kaohsiung Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SON KMU
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups: intervention (n=40) and contrast (n=40). Both groups received post-stroke usual care. The intervention group received an 8-week transitional care model for stroke patients, which included comprehensive discharge planning and home follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional care model (Experimental): In-hospital assessments, video-based stroke education, home visits, and weekly telephone follow-up
  Interventions: Behavioral: Transitional care model
- Post-stroke usual care (No Intervention): Treatment as usual after discharged home

INTERVENTIONS:
Behavioral: Transitional care model — In-hospital assessments, video-based stroke education, home visits, and weekly telephone follow-up
  Arms: Transitional care model

SUMMARY:
Patients with stroke benefitted from superior improvements in physical function, particularly when performing activities of daily living, fewer visits to the emergency room, less depression symptoms, and improved health-related quality of life thanks to transitional model care. Despite widespread implementation of transitional care for stroke patients, intervention effectiveness remains inconclusive, and another concern with transitional care for patients is the scarcity of effects on specific findings.

DETAILED DESCRIPTION:
A stroke may be a profound and life-changing occurrence for both the survivors and those who care for them, mandating participation in the adaptation and reinvention of a new post-stroke lifestyle that is sometimes unpredictable and temperamental. The sudden onset of a stroke and its accompanying treatment in an acute hospital setting can be distressing for both patients and caregivers. Admission after stroke may have a profound impact as patients and their caregiver start to understand the effects of the occurrence, which is scary, puzzling, and stressful. Nonetheless, adjusting to situations or life after a stroke might be made easier by implementing relevant and timely strategies throughout hospitalization, discharge, and the post-discharge period. Both populations, stroke patients and caregivers, may have unmet needs once the patients are discharged at home, such as communication, recovery plan and process, medicine, emotional needs, and stroke information, as well as social involvement. To address unmet needs after discharge from the hospital to a variety of settings, such transitional care is recommended to tackle the adverse outcomes.One of the widely used transitional care models is TCM, which was developed at the University of Pennsylvania under the direction of a nurse and was then made available to patients who were elderly at risk of poor outcomes and suffering from chronic illnesses including stroke patients. Incorporated into the model, TCM were developed to meet the needs that arose during hospitalization and to provide continuity of care for patients, including those with stroke, who were unable to receive it after their acute illness treatment

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old, being admitted in neurology department for at least 24 to 48 hours,
* Not having cognitive impairment as measured by the Montreal cognitive assessment (score ≥ 23),
* Being able to communicate in Indonesia, having the ability to provide informed consent,
* Being willing to participate in this study during hospitalization and 8 weeks after hospital discharge

Exclusion Criteria:

* Have potentially biased information, such as being unable to provide informed consent due to cognitive impairment,
* Having major speech and language problems or aphasia that prevent them from participating in the study,
* Having serious psychiatric disorders or other with terminal disease requiring active treatment, and
* Being discharged to a nursing home or welfare institution.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | Baseline, at week 4 intervention, and immediately post-intervention at week 8
  Self-efficacy has been proposed as an important determinant of the adaptation process in people who have had a stroke. The Indonesian version of Stroke Self-Efficacy Questionnaire (SSEQ-I) will be used in this study to assess participants' beliefs in their ability to perform and manage daily activities following a stroke. Participants rate their confidence in their ability to complete each of the 13 items on a 10-point scale, with 0 representing not at all confident and 10 representing very confident. Higher score indicates a higher level of self-efficacy (range 0-130).
Activities of daily living | Baseline, at week 4 intervention, and immediately post-intervention at week 8
  The ability to perform ADLs independently is a short-term rehabilitation goal during stroke recovery. The Indonesian version of the Modified Barthel Index (MBI-I) will be used to assess behavior related to activities of daily living in stroke patients or patients with other disabling conditions. The ten functional domains (activities) covered by this questionnaire include bowel and bladder control, grooming assistance, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing. Each item is graded on a scale of 0 to a maximum of 15. A total item score of less than or equal to 20 indicates total dependence, 21-60 severe dependence, 61-90 moderate dependence, 91-99 slight dependence and a total 100 indicates independence.

SECONDARY OUTCOMES:
Instrumental activities of daily living | Baseline, at week 4 intervention, and immediately post-intervention at week 8
  The Lawton IADL-Indonesian Version will be used to assess engagement in more complex activities in stroke patients. Each item is graded on a 2-point scale. The total score can range between 0 and 8. A total score is obtained by adding the items and normalizing to 8 for high function or independence for woman and 5 for man. For women, a score of 0 indicates total dependence or low function, 1-7 dependence or mild to moderate function, and a total 8 indicates independence or high function. For men, a score of 0 indicates total dependence or low function, 1-4 dependence or mild to moderate function, and a total 5 indicates independence or high function.
Depression symptoms | Baseline, at week 4 intervention, and immediately post-intervention at week 8
  Depression symptoms following a stroke covers roughly one-third of stroke survivors at any given time after the stroke. The Indonesian version of Geriatric Depression Scale (GDS), will be used to assess depression in stroke patients. Each item with 15 questions was scored on a 2-point scale (0 = "no," 1 = "yes"). Scores between 0 and 4 are considered normal, scores between 5-8, 9 to 11, and 12 to 15 indicate mild, moderate, and severe depression (range 0-15).
Quality of life in stroke patients | Baseline, at week 4 intervention, and immediately post-intervention at week 8
  The 26-item Indonesian version of World Health Organization Quality of Life-BREF (WHOQoL-BREF) will be used to assess the quality of life of stroke patients. This questionnaire comprises on four dimensions including physical health, psychological health, social relationships, and environmental health. Each dimension had five Likert response options, which were recoded into scores ranging from 0 to 4, with 0 being "never" and 4 being "always". Higher score indicates more severe of frequent problems or lower level of quality of life (range 0-104).

CONTACTS AND LOCATIONS:
Overall Officials: Bih-O Lee, Professor, Study Chair — Kaohsiung Medical University
Locations (1):
- RSUD Prof. Dr. W Z Johannes Kupang, Kupang, Indonesia

IPD SHARING:
Plan to Share IPD: No